CLINICAL TRIAL: NCT00599495
Title: Allogeneic Stem Cell Transplantation From Unrelated Donors After Dose-reduced Intensity Conditioning Regimen for Patients With Multiple Myeloma and Relapse After Autologous Stem Cell Transplantation: A Phase II-study
Brief Title: Matched Unrelated Donor Stem Cell Transplantation (MUD-SCT) After Dose-reduced Conditioning for Patients With Multiple Myeloma and Relapse After Autologous SCT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EBMT MUDRIC-MM
Record Dates: First submitted 2008-01-11; First posted 2008-01-23 (Estimated); Last update posted 2022-09-02 (Actual); Status verified 2022-09

CONDITIONS: Multiple Myeloma
Keywords: Hematopoietic Stem Cell Transplantation; Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: allogeneic HSCT — dose-reduced conditioning regimen

SUMMARY:
The purpose of this study is to determine whether a reduced intensity conditioning regimen followed by allogeneic stem cell transplantation from unrelated donors is a feasible and effective treatment for patients with multiple myeloma who failed a previous autologous stem cell transplantation.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether a reduced intensity conditioning regimen followed by allogeneic stem cell transplantation from unrelated donors is a feasible and effective treatment for patients with multiple myeloma who failed a previous autologous stem cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Multiple Myeloma stage II or III acc. to Salmon and Durie (chemosensitive or refractory) and relapse or progression after high dose chemotherapy with autologous stem cell support
* Age 18-60 years
* ECOG-performance status 0-1
* Availability of a HLA-compatible unrelated donor (HLA-A, -B, -DRB1, -DQB1)

Exclusion Criteria:

* Serious concomitant medical disease that would limit life span or ability to tolerate chemotherapy
* Severe cardiac failure (ejection fraction < 40%)
* Severe impairment of renal function (Creatinine clearance < 50ml/min)
* Severe impairment of liver function (bilirubine > 2 fold of upper limits of normal)
* Pregnant or lactating women
* Other major organ or system dysfunctions(GI, neurological, psychiatric dysfunctions that would impair tolerance of chemotherapy or prolonged haematological recovery)
* Positivity for HIV

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2002-11; Primary Completion 2009-08 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Engraftment, chimerism, toxicity, non-relapse mortality | Follow-up until day +1095

SECONDARY OUTCOMES:
Evaluation of response/GvHD/ infectious complications/ disease-free survival, Prognostic impact of cytogenetic, Evaluation of incidence and prognostic impact of molecular remission in patients with clinically complete remission. | Follow-up until day +1095

CONTACTS AND LOCATIONS:
Overall Officials: Nicolaus Kroeger, Prof. Dr., Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- University Medical Center Hamburg-Eppendorf, Hamburg, Germany

REFERENCES:
- [Result] Kroger N, Shimoni A, Schilling G, Schwerdtfeger R, Bornhauser M, Nagler A, Zander AR, Heinzelmann M, Brand R, Gahrton G, Morris C, Niederwieser D, de Witte T. Unrelated stem cell transplantation after reduced intensity conditioning for patients with multiple myeloma relapsing after autologous transplantation. Br J Haematol. 2010 Jan;148(2):323-31. doi: 10.1111/j.1365-2141.2009.07984.x. Epub 2009 Nov 12. PMID 19912215